CLINICAL TRIAL: NCT05491707
Title: Effect of Music on Patients' Anxiety During Lower Limb Arthroplasty Procedures Under Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Samantha Ballard, Principal investigator, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M210702; 202106_029 (Registry Identifier: The National Health Research Database)
Record Dates: First submitted 2022-08-01; First posted 2022-08-08 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Anxiety
Keywords: Music; Perioperative anxiety; Spinal anaesthesia; Lower limb arthroplasty
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: In this randomised controlled trial, patients will be identified on the arthroplasty lists. Criteria for inclusion will be determined at the pre-operative assessment. After enrolment, participants will be randomised into two groups in a 1:1 ratio, music (intervention group) and no music (control group). Randomisation will be done using a simple randomisation chart.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): Patients in the intervention group will receive music after the ASA monitors are applied. The music will be played at a self-selected volume, on Pro Bass Swagger Series Aux disposable earphones and will be played for the duration of the surgical procedure. The music will be played from an iPhone which will be placed in a plastic bag for infection control purposes. These patients will receive standard anaesthetic care.
  Interventions: Other: Music
- Control (No Intervention): The control group will not receive music. These patients will receive standard anaesthetic care.

INTERVENTIONS:
Other: Music — Patients will choose a genre of music from the following list; pop, gospel, classical, jazz, and soul, at the preoperative visit. This will be played on disposable ear phones at a self-selected volume for the duration of the surgical procedure.
  Arms: Music

SUMMARY:
The aim of this study is to compare the effect of listening to music, to a control group (no music), on peri-operative anxiety using the validated VAS-A, in patients undergoing lower limb arthroplasty procedures under spinal anaesthesia.

DETAILED DESCRIPTION:
Music is becoming an increasingly popular adjunct to traditional medical therapies. International studies have shown the numerous benefits of music in a medical setting. Music has been used effectively to decrease patients' anxiety under neuraxial anaesthesia for caesarean section. There is currently a lack of evidence supporting the use of music to reduce patients' anxiety under neuraxial anaesthesia for lower limb arthroplasty procedures. The worldwide growth of the ageing population has led to an increased demand for arthroplasty. It is imperative that the anaesthetic technique used for this procedure is both safe and is associated with high levels of patient satisfaction. The purpose of this study is to compare the effect of music, to a control, on peri-operative anxiety in patients undergoing lower limb arthroplasty procedures under spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* all patients, aged 18 years and older,
* American Society of Anaesthesiologists (ASA) class I, II or III,
* patients undergoing primary hip or knee arthroplasty surgery under spinal anaesthesia,
* patients with the mental capacity to consent to the study.

Exclusion Criteria:

* patients with significant visual or hearing loss,
* patients with any contra-indications to spinal anaesthesia,
* patients with any contra-indications to moderate sedation including moderate to severe obstructive sleep apnoea (indicated by a "STOPBANG" score of 5-8) (46),
* patients with pre-existing diagnosed anxiety disorders or other serious mental disturbances,
* revision arthroplasty (this may require deviation from the standardised anaesthetic technique used for this trial),
* anxious patients who cannot be reassured and require additional anxiolytic agents.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Describe the pre-operative anxiety scores measured by the visual analogue scale for anxiety | Pre-operative visit (T1)
  Describe the pre-operative anxiety scores measured by the visual analogue scale for anxiety in both the intervention and the control group. The minimum score on this scale is zero and the maximum score is ten. Zero indicates that the patients have no anxiety and ten indicates that the patient is extremely anxious.
Describe and compare the change in anxiety scores, on the visual analogue scale for anxiety, at the pre-operative visit (T1) and at skin incision (T3) in the control group. | Pre-operatively and skin incision
  Describe and compare the change anxiety scores, visual analogue scale for anxiety, at the pre-operative visit (T1) and at skin incision (T3) in the control group. The minimum score on this scale is zero and the maximum score is ten. Zero indicates that the patients have no anxiety and ten indicates that the patient is extremely anxious.
Describe and compare the change in anxiety scores, on the visual analogue scale for anxiety, at the pre-operative visit (T1) and at skin incision (T3) in the music group. | Pre-operatively and skin incision.
  Describe and compare the change in anxiety scores, on the visual analogue scale for anxiety, at the pre-operative visit (T1) and at skin incision (T3) in the music group. The minimum score on this scale is zero and the maximum score is ten. Zero indicates that the patients have no anxiety and ten indicates that the patient is extremely anxious.
Describe and compare the change in anxiety scores, on the visual analogue scale for anxiety, at each time point (T1-T4) between the control group and the music group. | Pre-operatively, prior to surgery, at skin incision and immediately after surgery.
  Describe and compare the change in anxiety scores, on the visual analogue scale for anxiety, at each time point (T1-T4) between the control group and the music group. The minimum score on this scale is zero and the maximum score is ten. Zero indicates that the patients have no anxiety and ten indicates that the patient is extremely anxious.

SECONDARY OUTCOMES:
Describe the difference in the anxiety scores, on the visual analogue scale for anxiety, between male and female patients. | Pre-operatively, prior to surgery, at skin incision and immediately after surgery.
  Describe the difference in the anxiety scores, on the visual analogue scale for anxiety, between male and female patients. The minimum score on this scale is zero and the maximum score is ten. Zero indicates that the patients have no anxiety and ten indicates that the patient is extremely anxious.
Describe the difference in anxiety scores, on the visual analogue scale for anxiety, between knee and hip arthroplasty. | Pre-operatively, prior to surgery, at skin incision and immediately after surgery.
  Describe the difference in anxiety scores, on the visual analogue scale for anxiety, between knee and hip arthroplasty. The minimum score on this scale is zero and the maximum score is ten. Zero indicates that the patients have no anxiety and ten indicates that the patient is extremely anxious.
Describe and compare the total propofol dose between the two groups. | Immediately after surgery
  Describe and compare the total propofol dose between the two groups.
Describe patient satisfaction, assessed by a questionnaire, in the intervention group. | Immediately after surgery
  Describe patient satisfaction, assessed by a questionnaire, in the intervention group. The questionnaire consists of five questions which patients will answer as either not at all, maybe, completely. The questions are: 1) Did the patient feel that the music decreased their anxiety? 2) Did the patient feel that the music provided calmness? 3) 3) Did the patient feel that they experienced less pain? 4) Would they request music again if coming for a similar procedure? 5) Would they recommend music to friends and family?

CONTACTS AND LOCATIONS:
Overall Officials: Samantha A Ballard, MBBCH, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Chris Hani Baragwanath Academic hospital, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification will be shared
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researches who provide a methodologically sound proposal.